CLINICAL TRIAL: NCT05094544
Title: Pre-Operative Immuno-Modulatory SBRT (POIMS Trial): A Pilot Trial in Early Stage NSCLC
Acronym: POIMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Shalina Gupta-Burt, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2020-POIMS-Lung
Record Dates: First submitted 2021-09-01; First posted 2021-10-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2022-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; SBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-ablative SBRT (Experimental): Non-ablative SBRT (800 cGy X 3 fractions) given 5-7 days preoperatively in selected patients with stage I-II NSCLC
  Interventions: Radiation: Non-ablative SBRT

INTERVENTIONS:
Radiation: Non-ablative SBRT — Non-ablative SBRT (800 cGy X 3 fractions) given 5-7 days preoperatively in selected patients with stage I-II NSCLC

SUMMARY:
The current proposal is structured as a pilot trial to evaluate the impact of non-ablative SBRT (800 cGy X 3 fractions) as an immunomodulatory mechanism in patients with early stage NSCLC who are surgical candidates. Tumor, normal tissue and blood specimens will be analyzed for immunomodulatory changes including phenotypic changes in tumor cell surface marker expression, tumor and normal tissue microenvironment and gene expression profiles, serum/blood immune profile changes, and circulating tumor cell immunophenotypic and gene expression alterations.

Published literature showed that cytotoxic doses of XRT may not elicit a clinically meaningful alteration in the immune profile. Further, studies using an animal model have concluded a fractionated regimen induces a greater abscopal effect than single dose radiation. Furthermore, research has shown a regimen of 800 cGy X 3 fractions yielded the most significant changes in the immune profile compared to 2000 cGy X 1 or 600 cGy X 5.

The immune response within the tumor milieu is a complex dynamic process with an interplay among lymphocyte subsets, antigen presenting cells/dendritic cells, macrophages, and tumor cells. The interactions between the various components is orchestrated by a variety of extracellular and intracellular signaling pathways involving ligand and cell surface expression, cytokine release, and activation or inhibition of a variety of T cell subsets. In order to comprehensively define the immunomodulatory effect of three fractions of 800 cGy on the primary tumor, the investigators will analyze the following: tumor cell surface phenotype, tumor microenvironment immune profile and gene expression profile, T cell repertoire changes in tumor tissue and peripheral blood, and circulating tumor cell phenotype and gene expression profiles. Each of these components has been shown to be impacted by radiation in either a cell culture or animal model systems. By characterizing, quantitating and defining these changes related to three fractions of 800 cGy, it will directly provide important insights to inform rational uses of XRT and immunotherapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-II NSCLC
* Adequate diagnostic biopsy tissue to allow pre-SBRT tumor analysis
* Candidate for oncologic surgery (lobectomy or sub lobar resection) for the lung cancer
* Lesion located peripherally, ≥ 2 cm from bronchial margin, and 1 cm from visceral pleura, with location deemed acceptable by cardio-thoracic surgeon for resection.
* Adequate pulmonary function test results

Exclusion Criteria:

* Prior history of lung/chest wall surgery
* Prior chest radiation
* Prior immunotherapy
* History of autoimmune disease
* Currently using immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Changes in tumor T cell repertoire following pre and post SBRT | through study completion, an average of 18 months
  Pre and post study intervention biopsy tissue comparison

SECONDARY OUTCOMES:
The impact of pre-surgical non-ablative SBRT on peri- and post-operative surgical complication rate | From Day of post-SBRT surgery through 6 month (± 2 months) post-operative follow up visit
  Medical Record Review Clavien-Dindo Classification system
Impact of SBRT on post-surgical wound healing complication rate assessed by CTCAE v5 | From Day of post-SBRT surgery through 6 month (± 2 months) post-operative follow up visit
  Medical record review General Thoracic Surgery Database.
Loco-regional control disease | From Day of enrollment through 36 month follow up visit
  Medical record review
  Loco-regional metastasisi
Metastasis-free survival | From Day of enrollment through 36 month follow up visit
  Medical record review
Overall survival | From Day of enrollment through 36 month follow up visit
  Medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Shalina Gupta-Burt, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

DOCUMENTS (2):
  • Study Protocol (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT05094544/Prot_000.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05094544/ICF_001.pdf